CLINICAL TRIAL: NCT07322380
Title: The FEDERATE-CAN Trial - FEasibility and aDoption of a scrEening pRogrAm for T1d rElatives in CANada
Brief Title: Feasibility and Adoption of a Screening Program for T1D Relatives in Canada
Acronym: FEDERATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2026-1340
Record Dates: First submitted 2025-12-11; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: screening; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Centralized approach (Active Comparator): Centralized approach managed and coordinated within the BETTER group based at IRCM (Montreal, Quebec), with standardized processes and integrated care pathways. In this approach, scheduling processes and data collection (clinical visits, laboratory analysis, questionnaires) will be handled by the research team. Participants' healthcare professional will be notified (by postal service and/or email if available)
  Interventions: Behavioral: Monitoring
- Decentralized approach (Active Comparator): In this approach, participants will be monitored by their preferred HCP according to consensus-based guidelines for monitoring pre-clinical T1D which will be communicated to both participants and HCPs. Therefore, follow-up and monitoring will be at the discretion of the HCP. However, regular contacts by the research team according to T1D stages will ensure the actual follow-up received.
  Interventions: Behavioral: Monitoring

INTERVENTIONS:
Behavioral: Monitoring — A semi-annual clinical visit (either by medical or trained staff) will be conducted to collect various data: IAb assessment, HbA1c measure, fasting blood glucose, glucose monitoring and information about eating habits, mental health, menstrual cycle, physical activity.

SUMMARY:
The aim of this study will be to evaluate the feasibility of an autoantibody-based type 1 diabetes screening program for first degree relatives of people living with type 1 diabetes within the province of Quebec. Feasibility of follow-up strategies of "at-risk" individuals will also be assessed.

This project will be divided into two phases, with the aim to evaluate:

1. The feasibility of a IAb (islet antibody)-based screening process for first degree relatives of people living with type 1 diabetes (T1D).
2. The feasibility of two approaches for follow-up monitoring in case of positive screening: centralized (within the organization) and decentralized approach (relying on individuals' healthcare providers), in the Quebec province setting.

Participants will come to the laboratory for blood sample collection, medical history and genetic risk score assessment, as well as anthropometric and cutaneous advanced glycated end (AGE) products measurements. A series of questionnaires will be completed.

After screening results are obtained (i.e., presence or absence of IAbs), a virtual visit will be conducted to communicate results to participants.

A positive result for IAb will warrant a second test for confirmation , using WBD within 3 months of initial screening.

After IAb positivity confirmation, participants will be invited to participate in phase 2 of this project (monitoring). Participants will be given the opportunity to select either a centralized or decentralized path for study monitoring.

Follow-up will be dependent of the stage of T1D:

* Participants in pre-stage 1 or stage 1 (2 or more positive IAbs without dysglycemia) T1D will receive a follow-up phone call six months after the initial screening.
* Participants in stage 2 (2 or more positive IAbs with dysglycemia) will be contacted one month after screening.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥18 years old living in the Québec province
* Having a FDR living with T1D (parents, siblings or offspring)
* Willing to adhere to follow-up care if screened positive

Exclusion Criteria:

* Having a diagnosis of T1D
* Pregnancy (ongoing or current attempt to become pregnant)
* Current or future expected use of glucocorticoid medication (except low stable dose and inhaled steroids and stable adrenal insufficiency treatment e.g., Cortef®) or any systemic immunosuppressive agents
* Planned or recent (< 6 weeks) monoclonal antibodies treatment, immunoglobulin perfusions or plasmapheresis.
* Other serious medical illness likely to interfere with study participation or with the ability to complete the study by the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of screening and monitoring outcomes | Through study completion for positive screened participants: 3 years
  Percentage of conversion of eligible participants to consent to participating in the study

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, M.D. Ph.D, Principal Investigator — Institut de recherches cliniques de Montréal

IPD SHARING:
Plan to Share IPD: No